CLINICAL TRIAL: NCT06840782
Title: First-line Immunotherapy-based Standard of Care and Local Ablative Treatments for Oligometastatic Non-small Cell Lung Cancer Patients: a Randomized, Multicentre, Open-label Phase III Study
Brief Title: First-line Immunotherapy-based Standard of Care and Local Ablative Treatments for Oligometastatic Non-small Cell Lung Cancer Patients.
Acronym: OliGRAIL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-503326-39-00; 2023/3729 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-01-16; First posted 2025-02-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Oligometastatic Non-small Cell Lung Cancer (NSCLC)
Keywords: Local ablative treatments; First-line immunotherapy; SBRT; Interventional radiology; Minimally invasive surgery
MeSH Terms: interventions — Minimally Invasive Surgical Procedures; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: RLT + SoC-based immunotherapy (+/- chemotherapy) (Experimental): RLT of all metastatic sites should be administered within 3 months after randomization and should not delay SoC-based immunotherapy administration.
  Interventions: Radiation: Radical local treatment; Drug: SoC-based immunotherapy (+/- chemotherapy)
- Control arm: SoC-based immunotherapy (+/- chemotherapy) (Active Comparator): SoC-based immunotherapy (+/- chemotherapy) will be administered every 3 weeks
  Interventions: Drug: SoC-based immunotherapy (+/- chemotherapy)

INTERVENTIONS:
Radiation: Radical local treatment — RLT of all metastatic sites. The possible RLT options will be SBRT, interventional radiology and/or minimally invasive surgery. Depending on the metastatic site, access and patient condition, the best RLT should be initially discussed in a case-to-case basis at the local multidisciplinary board (MTB).
  The primary tumour and initially invaded lymph nodes should be treated during the maintenance phase. Curative-intent approach modalities (e.g. hypofractionated intensity-modulated thoracic radiation therapy or surgery) should be discussed at the local MTB.
  Other Names: SBRT; Interventional radiology; Minimally invasive surgery
  Arms: Experimental arm: RLT + SoC-based immunotherapy (+/- chemotherapy)
Drug: SoC-based immunotherapy (+/- chemotherapy) — Current French SoC will be used. Main SoC-based immunotherapy includes:
  * Platinum-based chemotherapy combined with an anti PD-1 immunotherapy (pembrolizumab). Pemetrexed-platinum combinations may be used in non- squamous carcinoma, while paclitaxel-platinum combination is favoured in squamous carcinoma.
  * Anti PD-1 monotherapy if PD-L1 ≥ 50% is a possible alternative (pembrolizumab or atezolizumab or cemiplimab).
  Other alternatives include nivolumab-ipilimumab-chemotherapy or durvalumab-tremelimumab-chemotherapy association. Bevacizumab is not allowed given possible interactions with RLT.
  Maintenance/Immunotherapy alone will be pursued at the investigator's discretion according to the standard procedures (toxicity, progression, choice of the patient...).

SUMMARY:
First-line immunotherapy-based standard of care and local ablative treatments for oligometastatic non-small cell lung cancer patients: a randomized, multicentre, open-label phase III study

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced synchronous oligometastatic stage IV NSCLC.
* NSCLC patients eligible first line immunotherapy-based SoC according to the European Marketing Authorization.
* PDL1 status available.
* Metastases eligible to RLT according to the local multidisciplinary board (MTB): ≤5cm each in CT scan, excluding primary tumour.
* Maximum 5 metastases in 3 organs (EORTC criteria), according to brain MRI and FDG-PET.
* Symptomatic lesions requiring urgent palliative radiation, is permitted prior to randomization. These treated lesions should be counted towards the total number of metastases at the time of enrolment.
* Clinically required brain metastases (BM) ablation (surgery and/or SBRT) is permitted and BM count within the total number of 5 lesions. The patient would then be randomized to treatment of their extracranial disease.
* Acceptable organ function for RLT.
* ECOG performance status (PS) 0-1.
* Measurable lesions according to RECIST V1.1 on standard imaging.
* Patient aged 18 or more.
* Woman of childbearing potential must agree to use adequate contraception (implant type, vaginal ring, contraceptive pill, contraceptive patch, Intrauterine Device (IUD), etc.) for the duration of study participation and up to 6 months after completing treatment/therapy, in addition, male partners use a condom during this same period. Male patients must agree to use condom for the duration of study participation and up to 6 months after completing treatment/therapy.
* Patients affiliated to the social security system.
* Patient should understand, sign, and date the informed consent form written in French prior to any protocol-specific procedures performed.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

* Non-squamous NSCLC with targetable tumour mutations and approved first line targeted therapy (such as EGFR, ALK and ROS1).
* Metastases not eligible to RLT: e.g. brainstem or diffuse serosal metastases (meningeal, pericardial, pleural, peritoneal, mesenteric) or that invades the gastrointestinal tract.
* Brain metastases only, without extra-cerebral metastases.
* Uncontrolled severe comorbidity, symptomatic interstitial lung disease or active infection.
* Prior therapy with T-cell costimulation or immune checkpoint-targeted agents within 1 year.
* Uncontrolled concomitant (<1-year) malignancy except adequately treated basal or squamous cell carcinoma of the skin, or in-situ carcinoma of any organ or in-situ melanoma of the skin.
* Persons deprived of liberty by judicial or administrative decision.
* Persons subject to a legal protection measure (guardianship, curatorship, safeguard of justice).
* Persons not affiliated to a social security system or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS). | From date of randomization up to two years after the randomization of the last patient or documented death.
  Time from randomization to the date of documented death from any cause or last follow-up.

SECONDARY OUTCOMES:
Progression-free survival (PFS) according to RECIST 1.1. | From date of randomization up to two years after the randomization of the last patient or documented death.
  Time between the randomization date and the date of observation of a progression of the disease according to RECIST 1.1 or death of the patient (all causes combined) or date of last follow-up if the patient is alive without progression or lost to follow up.
immune Progression-free survival (iPFS) according to iRECIST. | From date of randomization up to two years after the randomization of the last patient or documented death.
  Time between the randomization date and the date of observation of an progression of the disease according to iRECIST 1.1 or death of the patient (all causes combined) or date of last follow-up if the patient is alive without progression or lost to follow up.
Number of side effects measured by CTCAE V.5. | From date of randomization up to two years after the randomization of the last patient or documented death.
  Acute/ late adverse events graded by CTCAE v5 (toxic death and serious adverse events) and their imputability to treatment.
EORTC Quality of Life Questionnaire-C30 (EORTC QLQ-C30). | From date of randomization up to 24 months after the last patient included in the study, until the date of first documented progression or date of death from any cause, whichever come first.
  The EORTC Quality of Life Questionnaire-C30 (EORTC QLQ-C30) contains 30 questions and assesses the quality of life of oncological patients multidimensionally over 10 subscales. All sub-scales and the 6 individual items have a score range from 0 to 100 points. A higher score represents better function and a higher quality of life. In the symptom subscale, however, a higher score represents a higher level of symptoms or problems.
EORTC Quality of Life Questionnaire Lung Cancer-specific-13 (QLQ-LC-13). | From date of randomization up to 24 months after the last patient included in the study, until the date of first documented progression or date of death from any cause, whichever come first.
  EORTC Quality of Life Questionnaire Lung Cancer-specific-13 (QLQ-LC-13) is a specific companion module used in conjunction with the EORTC QLQ-C30 and specifically developed for patients with Lung Cancer, and reliable in LC speciﬁc Qol assessment. The EORTC QLQ-LC13 comprises 13 item that measure lung cancer-related symptoms. Each items use the same 1-to-4 verbal response scale as the QLQ-C30 items, and domain scores are also transformed to a 0-to-100 metric. A higher score represents better function and a higher quality of life.
EuroQol-5D-5L Questionnaire (EQ-5D-5L). | From date of randomization up to 24 months after the last patient included in the study, until the date of first documented progression or date of death from any cause, whichever come first.
  The EuroQol-5D-5L Questionnaire (EQ-5D-5L) descriptive system of 5 health dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Index scores range from -0.59 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0. Used alongside the EQ-5D, the EQ visual analog scale (VAS) is a 20 cm VAS "assessing your own health today" with endpoints labeled "Best imaginable health state" (100) and "Worst imaginable health state" (0).
Clearance of circulating tumour DNA (ctDNA). | At the randomization, then Week 6 and Month 4 after randomization.
  ctDNA assessed in plasma.
Economic evaluation. | From date of randomization up to 24 months after the last patient included in the study, until the date of first documented progression or date of death from any cause, whichever come first.
  Incremental cost per Quality-adjusted life year (QALY based on EQ-5D-5L measures), incremental net monetary benefit. Assess the cost-utility (cost per QALY) of RLT + immunotherapy-based SoC compared to immunotherapy-based SoC alone.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut de Radiothérapie du Sud de l'Oise, Creil, Hauts-de-France
  - Centre Sainte-Catherine, Avignon, Provence-Alpes-Côte d'Azur Region
  - Gustave Roussy, Villejuif, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No